CLINICAL TRIAL: NCT06202378
Title: A Multicenter, Randomized, Double Blind, Placebo Controlled Phase II Clinical Study to Evaluate the Safety and Efficacy of SHPL-49 Injection in the Treatment of Acute Ischemic Stroke
Brief Title: Safety and Efficacy of SHPL-49 Injection in Participants With Acute Ischemic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Hutchison Pharmaceuticals Limited (Industry)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHPL-Z003-201
Record Dates: First submitted 2023-12-28; First posted 2024-01-11 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SHPL-49 Injection，3 ampoules (Experimental): 1mL/ampoule
  Interventions: Drug: 3 ampoules of SHPL-49 Injection
- SHPL-49 Injection，6 ampoules (Experimental): 1mL/ampoule
  Interventions: Drug: 6 ampoules of SHPL-49 Injection
- Placebo (Placebo Comparator): 1mL/ampoule
  Interventions: Drug: 0.9% Sodium Chloride Injection

INTERVENTIONS:
Drug: 3 ampoules of SHPL-49 Injection — 3 ampoules of SHPL-49 Injection in 100 mL 0.9% sodium chloride will be administered as a 30-minute intravenous infusion and applied twice daily for 7 days.
  Arms: SHPL-49 Injection，3 ampoules
Drug: 6 ampoules of SHPL-49 Injection — 6 ampoules of SHPL-49 Injection in 100 mL 0.9% sodium chloride will be administered as a 30-minute intravenous infusion and applied twice daily for 7 days.
  Arms: SHPL-49 Injection，6 ampoules
Drug: 0.9% Sodium Chloride Injection — 100 mL 0.9% sodium chloride will be administered as a 30-minute intravenous infusion and applied twice daily for 7 days.
  Arms: Placebo

SUMMARY:
This study is designed to determine the safety and efficacy of SHPL-49 intravenous infusion for 7 consecutive days in the treatment of acute ischemic stroke subjects.

DETAILED DESCRIPTION:
Trial Objectives:

The primary objective of this study is to determine the effectiveness of different doses of SHPL-49 intravenous infusion for 7 consecutive days in the treatment of acute ischemic stroke subjects within 8h after onset.

The secondary objective is to determine the safety of different doses of SHPL-49 intravenous infusion for 7 consecutive days in the treatment of acute ischemic stroke subjects within 8h after onset.

Trial Design:

This study is a Phase II, multicenter, randomized, double Blind, placebo-Controlled design. Participants receive twice daily dosing for 7 consecutive days, or once on Days 1 and Day 8 and twice daily on Days 2 to Day 7, with each subject scheduled to receive 14 doses throughout the clinical trial. 270 Participants will be randomized 1:1:1 to SHPL-49 injection treated group (3 ampoules of SHPL-49 injections, Bis in die（BID）), SHPL-49 injection treated group (6 ampoules of SHPL-49 injections , BID) and placebo group (BID).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old (including upper and lower limits);
2. Clinically diagnosed as acute ischemic stroke according to the latest guidelines;
3. Patients with acute ischemic stroke who plan to receive or have received standard intravenous thrombolysis in hospital (this research center) within 8h after the onset of the disease;
4. Participants who have NIHSS ≥5 and ≤ 22 before thrombolysis;
5. Pre-stroke mRS Score ≤1;
6. Participants or legally authorized representatives who are able and willing to sign informed consent.

Exclusion Criteria:

1. Complicated with intracranial hemorrhagic diseases, including hemorrhagic stroke, epidural hematoma, intracranial hematoma, ventricular hemorrhage, subarachnoid hemorrhage, etc.;
2. Severe disturbance of consciousness: patients with NIHSS 1a consciousness level item score ≥2;
3. Cerebral Computed tomography (CT) or Magnetic resonance imaging (MRI) indicated a large anterior circulation cerebral infarction (ASPECT score < 6 or infarct area greater than 1/3 of the middle cerebral artery blood supply area);
4. Stroke with rapid improvement of symptoms before intravenous thrombolysis, or acute ischemic symptoms suspected to be caused by other causes;
5. Patients who are ready to receive or have receive intravascular therapy;
6. After the onset of the disease, drugs with neuroprotective effects have been applied in the instructions. Such as commercially available Edaravone, Edaravone and Dexborneol Concentrated Solution for Injection, Butylphthalide, Nimodipine, Ganglioside, Citicoline, Piracetam, Oxiracetam, Human Urinary Kallidinogenase, Cinepazide, Mouse Nerve Growth Factor For Injection, Cerebrolysin, Deproteinised Calf Blood Serum Injection, Deproteinised Calf Blood Extractives Injection, etc.;
7. Severe hypertension: systolic blood pressure ≥185mmHg or diastolic blood pressure ≥110mmHg after taking antihypertensive drugs before thrombolysis;
8. Severe renal insufficiency: serum creatinine >2 times the upper limit of normal or creatinine clearance (CLcr)< 30mL/min (Cockcroft-Gault formula), or other known severe renal insufficiency; (Note: Cockcroft-Gault formula: ① Male: CLcr (mL/min) = [140 - age (yrs)]× body weight (kg) / [0.814 × serum creatinine (μmol/L)]; (2) female: CLcr (mL/min) = {[140 - age (years old)] by weight (kg) / [0.814 x serum creatinine (μmol/L)]} x 0.85)
9. Severe liver function impairment: Alanine aminotransferase (ALT) or Aspartate aminotransferase(AST)>3 times the upper limit of normal, or other known liver diseases such as acute and chronic hepatitis, cirrhosis, etc.;
10. Patients with a heart function rating above Class II (according to the New York Heart Association (NYHA) heart function rating) or a history of congestive heart failure;
11. Patients with concurrent malignant tumors or undergoing anti-tumor therapy;
12. Allergic to experimental drugs or similar ingredients or materials used in imaging examinations;
13. Patients during pregnancy, breastfeeding or planning pregnancy;
14. Patients who have a history of epilepsy or have had seizure-like symptoms at the onset of stroke, or suffer from serious mental disorders, intellectual disabilities or dementia;
15. Suspected or confirmed alcohol dependence, or drinking more than 3 units (male) or 2 units (female) of alcohol within 24 hours prior to onset (1 unit =360 mL beer or 45 mL liquor with 40% alcohol or 150 mL wine);
16. Patients have participated in or are participating in another clinical study within the 3 months before singing informed consent;
17. Patients who are judged unsuitable for participation by the investigators in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2023-12-29 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS), with scores of 0-1 at Day 90 | 90±7 days
  Proportion of participants with mRS scores of 0-1 at Day 90

SECONDARY OUTCOMES:
Shift analysis/ Ordinal analysis | 90±7 days
  A shift of one or more categories to reduced functional dependence analyzed across the whole distribution of outcomes on the mRS at Day 90
Modified Rankin Scale (mRS), with scores of 0-1 at Day 30 | 30±3 days
  Proportion of participants with mRS Scores of 0-1 at Day 30
Modified Rankin Scale (mRS), with scores of 0-2 at Day 30 | 30±3 days
  Proportion of participants with mRS Scores of 0-2 at Day 30
Modified Rankin Scale (mRS), with scores of 0-2 at Day 90 | 90±7 days
  Proportion of participants with mRS Scores of 0-2 at Day 90
National Institute of Health stroke scale (NIHSS) on day 7or 8 | 7 days or 8 days
  The proportion of participants with NIHSS scores of 0-1 or with ≥4 point reduction from baseline on day 7 or 8 (after the completion of the final dose)
National Institute of Health stroke scale (NIHSS) at Day 14 or at discharge | 14±2 days
  The proportion of participants with NIHSS scores of 0 to 1 or with 4 points reduction from baseline on day 14 or at discharge
Barthel index (BI) at Day 30 | 30±3 days
  Proportion of participants with Barthel index ≥95 at Day 30
Barthel inde (BI) at Day 90 | 90±7 days
  Proportion of participants with BI ≥95 at Day 90
National Institute of Health stroke scale (NIHSS) at Day 14 or at discharge | 14±2 days or at discharge
  Changes in NIHSS scores from baseline at Day 14 or at discharge
Symptomatic intracranial hemorrhage | 22-36h after thrombolysis
  Symptomatic intracranial hemorrhage within 36h after thrombolysis (Safe Implementation of Thrombolysis in Stroke-Monitoring Study Criteria)
Mortality | 90±7 days
  Mortality over the 90-day study period
Serious adverse events | 90±7 days
  Serious adverse events over the 90-day study period
Adverse events | 90±7 days
  Adverse events over the 90-day study period
Changes in laboratory test indicators | 7 days or 8 days，14±2 days，90±7 days
  Changes in laboratory test indicators on day 7 or 8(at the end of the last dose), at Day 14 or at discharge, and at Day 90
Changes in vital signs before and after administration | 7 days or 8 days，14±2 days，90±7 days
  Changes in vital signs on day 7 or 8 (at the end of the last dose), at Day14 or at discharge , and at Day 90
12-lead electrocardiogram | 90±7 days
  Abnormal 12-lead electrocardiogram over the 90-day study period
Vital signs | 90±7 days
  Abnormal vital signs over the 90-day study period
Physical examination | 90±7 days
  Abnormal results of physical examination over the 90-day study period
Laboratory test indicators | 90±7 days
  Abnormal laboratory test indicators over the 90-day study period

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, master, Principal Investigator — Beijing Tiantan Hospital
Locations (16):
- China (16):
  - Beijing Tiantan Hosptial，Capital Medical University, Beijing, Beijing Municipality
  - Yuebei People's Hospital, Shaoguan, Guangdong
  - Hengshui People's Hospital, Hengshui, Hebei
  - Tangshan Workers' Hospital, Tangshan, Hebei
  - Nanshi Hospital of Nanyang, Nanyang, Henan
  - General Hospital of Pingmei Shenma Group, Pingdingshan, Henan
  - Keshiketeng Banner Traditional Chinese Medicine and Mongolian Medicine Hospital, Chifeng, Inner Mongolia
  - The First Hospital of Jilin University, Changchun, Jilin
  - Beipiao Central Hospital, Beipiao, Liaoning
  - Shenyang Medical College Affiliated Central Hospital, Shenyang, Liaoning
  - The First People's Hospital of Shenyang, Shenyang, Liaoning
  - Linyi People's Hospital, Linyi, Shandong
  - The First People's Hospital of Tancheng, Linyi, Shandong
  - Sinopharm Tongmei General Hospital, Datong, Shanxi
  - Linfen Central Hospital, Linfen, Shanxi
  - Linfen People's Hospital, Linfen, Shanxi